CLINICAL TRIAL: NCT00489567
Title: A Hospital-based Surveillance to Collect Prospective Data to Estimate the Disease Burden of Severe RV GE, Its Complications and Diversity of Co-circulating Rotavirus Strains in Children < 5 Years of Age in Sweden
Brief Title: Hospital-based Surveillance to Collect Prospective Data to Estimate the Disease Burden of Severe RV GE in Sweden
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Other Study IDs: 109551
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Rotavirus Gastroenteritis; Infections, Rotavirus
Keywords: Rotavirus gastroenteritis
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample, Blood sample

GROUPS / COHORTS (1):
- Group A: Children hospitalised with community-acquired severe RV GE and children acquiring nosocomial severe RV GE.
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection

SUMMARY:
This study aims to estimate the burden of RV GE. The study will focus on children hospitalized for severe RV GE, Children acquiring RV GE in the hospital and the household contacts of children hospitalized with RV GE. It is expected to enrol 500-600 subjects in the study. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from parent or guardian
* A male/ female child aged less than 5 years. On the day of fifth birthday the subject is not eligible for participation
* Hospitalised for acute GE
* Developed symptoms of acute GE 72 hours after hospitalisation
* Stool sample should be positive for the presence of rotavirus, which will be detected either by Vikia test or by ELISA

Inclusion criteria for household members:

* Family members including care-takers and sibling staying in the same house and who spend most of the nights (50%) with the sick child.
* Written permission from care-takers or siblings or their parents.

Exclusion Criteria:

- All children in the neonatal wards.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children < 5 years of age in Sweden
Sampling Method: Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence of severe rotavirus gastroenteritis (RV GE) and its associated complications in children < 5 years of age.

SECONDARY OUTCOMES:
To determine the gender, age of onset, severity of symptoms and underlying medical conditions in community and nosocomially acquired rotavirus infections
To check the incidence of RV antigenemia and viremia associated with severe RV GE and relate this to clinical symptoms and rate of complications in population under surveillance.
To estimate the incidence of liver involvement associated with RV GE and relate this to clinical symptoms in the population under surveillance.
To explore the possible role of anti-secretory factor in children with RV GE and relate this to clinical symptoms and rate of complications under surveillance.
To genotype the isolated rotavirus strains and evaluate a possible correlation to evolved antigenemia, liver involvement and complications in both nosocomially and community-acquired cases with infection of different strain

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline